CLINICAL TRIAL: NCT02581930
Title: A Phase 2 Study of Ibrutinib (PCI-32765) in Refractory Distant Metastatic Cutaneous Melanoma: Correlation of Biomarkers With Response and Resistance
Brief Title: Ibrutinib in Treating Patients With Refractory Metastatic Cutaneous Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-01744; NCI-2015-01744 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI9922; 9922 (Other: Duke University - Duke Cancer Institute LAO); 9922 (Other: CTEP); UM1CA186644 (NIH); UM1CA186686 (NIH); UM1CA186688 (NIH); UM1CA186689 (NIH); UM1CA186690 (NIH); UM1CA186691 (NIH); UM1CA186704 (NIH); UM1CA186709 (NIH); UM1CA186712 (NIH); UM1CA186716 (NIH); UM1CA186717 (NIH); NCT03427398 (obsolete NCT alias)
Record Dates: First submitted 2015-10-20; First posted 2015-10-21 (Estimated); Results first posted 2019-06-18 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Melanoma; Recurrent Cutaneous Melanoma; Stage IV Cutaneous Melanoma AJCC v6 and v7
MeSH Terms: conditions — Melanoma | interventions — ibrutinib; Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (ibrutinib) (Experimental): Patients receive ibrutinib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Other: Laboratory Biomarker Analysis; Other: Pharmacogenomic Study; Other: Pharmacological Study

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA 032765; CRA-032765; CRA032765; Imbruvica; PCI 32765; PCI-32765; PCI32765
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacogenomic Study — Correlative studies
  Other Names: PHARMACOGENOMIC
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies how well ibrutinib works in treating patients with stage IV melanoma of the skin that has not responded to previous treatment. Ibrutinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate rate of objective response (OR: complete response [CR] + partial response [PR]) to ibrutinib administered as single agent in patients with immune checkpoint inhibitor-refractory, or immune checkpoint inhibitor ineligible and mitogen-activated protein kinase (MAPK) inhibitor-refractory (if B-Raf proto-oncogene, serine/threonine kinase [BRAF]V600-mutant) or MAPK inhibitor-intolerant distant metastatic cutaneous melanoma.

SECONDARY OBJECTIVES:

I. Estimate progression-free survival (PFS) rate at 6 months after initiation of ibrutinib in patients with immune checkpoint inhibitor-refractory or immune checkpoint ineligible and MAPK inhibitor-refractory (if BRAFV600-mutant) or MAPK inhibitor-intolerant distant metastatic cutaneous melanoma.

II. Estimate overall survival (OS) after initiation of ibrutinib in patients with immune checkpoint inhibitor-refractory or immune checkpoint ineligible and MAPK inhibitor-refractory (if BRAFV600-mutant) or MAPK inhibitor-intolerant distant metastatic cutaneous melanoma.

III. Explore the association of ITK protein expression with OR and PFS.

TERTIARY OBJECTIVES:

I. Explore association between other putative targets of ibrutinib (e.g. Tec, ErbB4, Hck, Yes, BTK) in melanoma cells, as assessed by 2-color immunofluorescence (IF) in representative tissue sections obtained from pretreatment archived formalin-fixed paraffin-embedded (FFPE) tumor blocks or FFPE blocks obtained from fresh tissue biopsy from enrolled patients, with overall response (OR) and PFS.

II. Explore ibrutinib-mediated effect(s) on immune cell subsets associated with immunomodulation by performing multiparameter flow cytometric analysis in peripheral blood mononuclear cell (PBMC) obtained prior to treatment, on day 29 (i.e., predose day 1 of cycle 2) following initiation of treatment with ibrutinib, and at the time of disease progression (3 time points).

III. Determine pharmacokinetics (PK) of ibrutinib following daily dosing at 840 mg on day 8 of cycle 1 (Css).

OUTLINE:

Patients receive ibrutinib orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed melanoma of cutaneous primary; metastatic melanoma from unknown primary are allowed
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 10 mm (>= 1 cm) with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Stage IV disease
* If BRAFV600-mutant, documented refractory disease to at least one BRAF inhibitor (dabrafenib or vemurafenib) and/or a MEK inhibitor (trametinib or cobimetinib), defined as progression of measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST) criteria while on treatment; subjects with MAPK inhibitor-intolerance are eligible if they meet criteria
* Documented disease refractory to at least one PD1/PD-L1 inhibitor, defined as disease progression following at least 2 infusions of the same drug; radiographic disease progression will be documented by the institutional radiologist based on any radiographic evidence (magnetic resonance imaging [MRI], computed tomography [CT], positron emission tomography [PET], or other modalities, etc.) of disease progression on two separate radiographic scans assessment obtained at least 4 weeks apart; this minimum 4-week interval is required to define PD-1 inhibitor resistance based on imaging; alternatively, clinical disease progression may be documented on examination by the treating investigator
* Prior treatment-related toxicity resolved to =< grade 1 or baseline with the exception of alopecia and permanent grade =< 2 toxicities related to prior immune checkpoint inhibitor treatment (e.g. PD-1/PD-L1, CTLA-4, CD40, LAG3) treatment with the review and approval by the lead principal investigator (PI)
* Prior radiation allowed (no restriction on amount); measurable lesion(s) may not have been previously irradiated
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 3 months
* Hemoglobin >= 9.0 g/dL
* Absolute neutrophil count (ANC) > 1,500/uL
* Platelets > 100,000/uL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2 x upper limit of normal (ULN); =< 5 x ULN, if liver metastasis
* Total bilirubin =< 1.5 x ULN unless Gilbert's syndrome of disease infiltration of the liver is present
* Creatinine clearance estimated glomerular filtration rate (GFR) >= 30 mL/min/1.73 m^2 (Cockcroft-Gault)
* Patients with brain metastases are allowed provided that:

  * No leptomeningeal disease is present
  * Intracranial disease is controlled by prior local therapies (craniotomy, stereotactic radiosurgery, whole brain irradiation), as evidenced by brain MRI 4 weeks post treatment indicating no new intracranial disease
  * Stable or decreasing dose of steroids provided patient on =< 20 mg of prednisone or its equivalent daily
* Ibrutinib should be held at least 3 to 7 days pre- and post-surgery, depending upon the type of surgery and risk of bleeding
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 90 days after completion of ibrutinib administration; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 90 days after completion of ibrutinib administration
* Negative serum pregnancy test within 7 days of treatment initiation with ibrutinib in women of childbearing potential (WOCBP)
* Ability to swallow oral medications
* Patients with autoimmune disease requiring systemic corticosteroid treatment (and previously ineligible to receive systemic immunotherapies for melanoma) are allowed on condition that they do not receive more than 20 mg of daily dose methylprednisolone, prednisone, or its equivalent; this does not include autoimmune diseases caused by previous immunotherapy treatments for melanoma that require ongoing treatment with corticosteroids (e.g. autoimmune colitis or autoimmune hepatitis receiving corticosteroids)
* Willing to consent to allow access to known archival tumor tissue (NOTE: designated pathologist from participating site OR lead principal investigator must sign-off to ensure "sufficient" tumor should be available for support of tumor imaging studies [multi-color immunofluorescence])
* If archival tumor tissue from a metastatic melanoma lesion is unavailable OR designated pathologist from participating site cannot sign-off to ensure that "sufficient" tumor is available from existing archival tumor block for support of tumor imaging studies, patients must be willing to consent to undergo a biopsy to collect metastatic tumor tissue; collection of fresh biopsy tissue does not guarantee enrollment, unless the pathologist from the participating site signs-off that "sufficient" tumor has been collected
* Ability to understand and the willingness to sign a written informed consent document
* Subjects who are unable to tolerate BRAF inhibitor and/or MEK inhibitor therapy due to grade >= 2 toxicity (Common Terminology Criteria for Adverse Events [CTCAE] version [v]4.0) from these agents, irrespective of antitumor response, are eligible on condition that: (a) toxicities persisted despite change from doublet to singlet therapy (i.e. from concurrent BRAF inhibition plus MEK inhibition to BRAF inhibition alone), (b) toxicities are attributed to a class effect, and therefore switch from one drug to another is expected to induce the same type of toxicity (e.g. ocular toxicities or cardiac dysfunction from MEK inhibitor), (c) drug-specific toxicities that do not resolve with switch from one BRAF inhibitor to another (i.e. dabrafenib to vemurafenib, or vice versa), will be eligible for enrollment in 9922; in other words, patients will be allowed to enroll into the NCI9922 study despite lack of progression to MAPK inhibitor treatments, on condition that grade 2 or higher toxicities attributed to MAPK inhibitors resolve to grade 1, or less, at the time of study enrollment

Exclusion Criteria:

* Patients with melanoma of mucosal or ocular primary
* Patients who have had chemotherapy or immunotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) or radiotherapy within 2 weeks prior to cycle 1 day 1; patients who have had tyrosine kinase inhibitors (such as Braf or MEK inhibitors) within 15 days of cycle 1 day 1
* Patients who are receiving any other biologic, cytotoxic or investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ibrutinib (difficulty breathing, lip swelling, itching or rash)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant and breastfeeding women are excluded from this study; breastfeeding should be discontinued if the mother is treated with ibrutinib
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are eligible; unless the patient's cluster of differentiation (CD)4+ count is below the institutional lower limit of normal
* Uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenic purpura (ITP) resulting in (or as evidenced by) declining platelet or hemoglobin (Hgb) levels within the 4 weeks prior to first dose of study drug
* Presence of transfusion-dependent thrombocytopenia
* Need for daily corticosteroids at high doses (prednisone >= 20 mg daily, or an equivalent) is prohibited from 28 days prior to first dose and during treatment with ibrutinib; brief (up to 7 days) and episodic use of systemic corticosteroids for other general conditions (e.g. pre-medication for radiographic imaging due to intravenous [IV] contrast allergy, chronic obstructive pulmonary disease [COPD] exacerbation, poison ivy, etc.) is allowed
* Prior exposure to ibrutinib or other ITK inhibitors
* History of prior malignancy, with the exception of the following:

  * Non-melanoma skin cancers, non-invasive bladder cancer, and carcinoma in situ of the cervix
  * Prostate cancer not under active systemic treatment other than hormonal therapy and with documented undetectable prostate-specific antigen (PSA) (< 0.2 ng/mL)
  * Chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL) provided patient has isolated lymphocytosis (Rai stage O), and does not require systemic treatment (for "B" symptoms, Richter's transformation, lymphocyte doubling time [< 6 months], lymphadenopathy or hepatosplenomegaly)
  * Lymphoma of any type of hairy-cell leukemia provided patient is not on active systemic treatment and is in complete remission, as evidenced by PET/CT scans and bone marrow biopsies for at least 3 months
  * History of malignancy provided that patient has completed therapy and is free of disease for >= 2 years; if patient had other malignancy within the last 2 years from which he may have been completely cured by surgery alone, he may be considered to be enrolled on condition that the risk of development of distant metastatic disease based on American Joint Committee on Cancer (AJCC) staging system is less than 30%
* Currently active clinically significant cardiovascular disease, such as uncontrolled arrhythmia, congestive heart failure, any class 3 or 4 cardiac disease, as defined by the New York Heart Association Functional Classification, or history of myocardial infarction within 6 months prior to first dose with study drug
* Unable to swallow capsules, or disease significantly affecting gastrointestinal function and/or inhibiting small intestine absorption, such as malabsorption syndrome, resection of portions of small bowel larger than 3 feet, or poorly controlled inflammatory bowel disease affecting the small intestine
* Known serologic status reflecting active hepatitis B or C infection; patients that are hepatitis B core antibody positive, but antigen negative, will need a negative polymerase chain reaction (PCR) prior to enrollment (NOTE: hepatitis B antigen or PCR positive patients will be excluded)
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment
* Current life-threatening illness, medical condition, or organ system dysfunction, which, in the investigator's opinion, could compromise the patient's safety, or put the study at risk
* Received anticoagulation therapy with warfarin, or equivalent vitamin K antagonists, within the last 28 days prior to day 1 of ibrutinib; patients with familial coagulopathic diseases (e.g. hemophilia, von Willebrand disease) are also excluded; if applicable, subjects must discontinue fish oil and vitamin E supplements within 7 days prior to initiating ibrutinib therapy
* Subjects with known hepatic insufficiency (i.e. Child-Pugh score A [mild], Child-Pugh score B [moderate] or Child-Pugh score C [severe]) according to Child-Pugh criteria
* Subjects who received a strong cytochrome P450 (CYP) 3A inhibitor within 7 days prior to the first dose of ibrutinib or subjects who require continuous treatment with a strong CYP 450 3A inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-08-17 (Actual); Primary Completion 2018-02-10 (Actual); Study Completion 2026-03-17 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Stergios J Moschos, Principal Investigator — Duke University - Duke Cancer Institute LAO
Locations (13):
- United States (13):
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Washington University School of Medicine, St Louis, Missouri
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

REFERENCES:
- [Derived] Moschos SJ, Eroglu Z, Khushalani NI, Kendra KL, Ansstas G, In GK, Wang P, Liu G, Collichio FA, Googe PB, Carson CC, McKinnon K, Wang HH, Nikolaishvilli-Feinberg N, Ivanova A, Arrowood CC, Garrett-Mead N, Conway KC, Edmiston SN, Ollila DW, Serody JS, Thomas NE, Ivy SP, Agrawal L, Dees EC, Abbruzzese JL. Targeting the IL-2 inducible kinase in melanoma; a phase 2 study of ibrutinib in systemic treatment-refractory distant metastatic cutaneous melanoma: preclinical rationale, biology, and clinical activity (NCI9922). Melanoma Res. 2021 Apr 1;31(2):162-172. doi: 10.1097/CMR.0000000000000726. PMID 33661190

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of the recruitment period were 12/12/16-12/14/17 in medical clinic.
Period: Overall Study
Arm/Group | Treatment (Ibrutinib)
Started | 18
Completed | 16
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — patient declined further treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 18
Age, Continuous [Mean (Full Range); unit: years] | 60 [37 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Antitumor Response as Evaluated by Response Evaluation Criteria in Solid Tumors (RECIST) Criteria 1.1
Description: Antitumor response defined as the sum of complete response (CR) and partial response (PR). CR is the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm (<1 cm). PR is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 18
Participants | 0
Statistical Analysis 1: Comparison: Treatment (Ibrutinib); The primary comparison was between the response rate of an ineffective drug, such as investigators' choice chemotherapy (5%), and the response rate of ibrutinib; Test type: Other — Exact binomial test; p = 1.00, Exact binomial test, 1-sided — Significant if p-value is less than 0.1; Probability of response = 0.00 — Estimated as proportion of subjects with response

2. Secondary Outcome: Progression Free Survival
Description: Progression free survival (PFS) is defined as the duration of time from Day 1 of treatment to time of progression (based on clinical or radiographic grounds) or death as a result of any cause, whichever occurs first.
Time Frame: 1 year
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 18
months | 1.3 [0.2 to 5.5]

3. Secondary Outcome: Overall Survival
Description: Estimated using the Kaplan Meier method.
Time Frame: Duration of time from day 1 of treatment to death as a result of any cause, assessed up to 1 year
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 18
months | 6 [0.3 to 6.7]

4. Other Pre Specified Outcome: Expression Levels of ITK and Putative Targets of Ibrutinib (e.g. Tec, ErbB4, Hck, Yes, BTK)
Description: Assessed by IHC and 2-color IF and analyzed by Aperio imaging. Exploratory analysis will also be performed to assess the predictive ability of each tissue biomarker by fitting logistic model or Cox model with biomarker as a covariate. Antitumor response rate or PFS information will be used to investigate possible cut-points for the biomarker. Logistic regression analysis will be conducted to assess whether a profile of immune response in tumor biopsies (or in peripheral blood) can be developed that distinguishes patients who respond to treatment versus those who do not.
Time Frame: Up to 1 year
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change in Th1, Th2, and Various Immune Regulatory Cell Populations in Peripheral Blood Mononuclear Cells and Assessed by Flow Cytometry
Description: Will be assessed by comparisons using analysis of variance followed by paired t-test or other tests (Wilcoxon rank-sum test), if normality assumption is not satisfied even when data transformation is performed.
Time Frame: Baseline up to 1 year
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Pharmacokinetic Analysis on Ibrutinib Concentrations in Plasma Using WinNonlin
Description: The following parameters will be estimated: maximum concentration, time of maximum concentration, area under the concentration verses time curve, half-life, apparent clearance, apparent volume of distribution.
Time Frame: Pre-dose on days 1 and day 8 of course 1 and post-dose, 0.5, 1, 2, 4, 6, and 24 hours on day 8 of course 1
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Treatment (Ibrutinib)
All-Cause Mortality (participants affected / at risk) | 15/18
Serious Adverse Events (participants affected / at risk) | 9/18
Other Adverse Events (participants affected / at risk) | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Ibrutinib) (N=18)
sepsis (Infections and infestations) | 1
cytokine release syncrome (Immune system disorders) | 1
constipation (Gastrointestinal disorders) | 1
hyponatremia (Renal and urinary disorders) | 4
hypotension (Vascular disorders) | 1
hypertension (Vascular disorders) | 1
dehydration (Metabolism and nutrition disorders) | 1
decreased lymphocyte count (Blood and lymphatic system disorders) | 1
pneumonia (Infections and infestations) | 1
anemia (Blood and lymphatic system disorders) | 1
hypoalbuminemia (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Ibrutinib) (N=18)
anemia (Blood and lymphatic system disorders) | 7
anorexia (Gastrointestinal disorders) | 10
fatigue (General disorders) | 10
nausea (Gastrointestinal disorders) | 5
diarrhea (Gastrointestinal disorders) | 4
decreased neutrophil count (Blood and lymphatic system disorders) | 1
decreased platelet count (Blood and lymphatic system disorders) | 1
decreased WBC (Blood and lymphatic system disorders) | 1
increased neutrophil count (Blood and lymphatic system disorders) | 1
increased WBC count (Blood and lymphatic system disorders) | 1
vomiting (Gastrointestinal disorders) | 4
hypoalbuminemia (Hepatobiliary disorders) | 3
hypomagnesemia (Metabolism and nutrition disorders) | 2
hypophosphatemia (Metabolism and nutrition disorders) | 1
hyponatremia (Metabolism and nutrition disorders) | 1
hypertension (Cardiac disorders) | 2
palpitations (Cardiac disorders) | 1
constipation (Gastrointestinal disorders) | 1
headaches (Nervous system disorders) | 2
fever (General disorders) | 3
chills (General disorders) | 2
dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
oral mucositis (Gastrointestinal disorders) | 2
hypokalemia (Metabolism and nutrition disorders) | 1
hypocalcemia (Metabolism and nutrition disorders) | 1
dysgeusia (Gastrointestinal disorders) | 2
rash (Skin and subcutaneous tissue disorders) | 4
bruising (Skin and subcutaneous tissue disorders) | 2
diziness (Nervous system disorders) | 2
dehydration (Metabolism and nutrition disorders) | 1
hematuria (Renal and urinary disorders) | 1
proteinuria (Renal and urinary disorders) | 1
limb edema (Musculoskeletal and connective tissue disorders) | 2
blurry vision (Eye disorders) | 1
eye redness (Eye disorders) | 1
anxiety (Nervous system disorders) | 1
lethargy (General disorders) | 1
flushing (Skin and subcutaneous tissue disorders) | 1
pruritus (Skin and subcutaneous tissue disorders) | 1
sinus tachycardia (Cardiac disorders) | 1
AlPhos increased (Metabolism and nutrition disorders) | 1
Bilirubin increased (Hepatobiliary disorders) | 1
tremor (Nervous system disorders) | 2
insomnia (Nervous system disorders) | 1
dysphagia (Gastrointestinal disorders) | 1
hiccups (Gastrointestinal disorders) | 1
restless legs (Musculoskeletal and connective tissue disorders) | 1
joint effusion (Musculoskeletal and connective tissue disorders) | 1
hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
tooth infection (Infections and infestations) | 1
urinary tract infection (Infections and infestations) | 1
facial edema (Musculoskeletal and connective tissue disorders) | 1
trunk edema (Musculoskeletal and connective tissue disorders) | 1
pain (General disorders) | 2
abdominal pain (General disorders) | 1
flank pain (General disorders) | 1
sinusitis (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT02581930/Prot_SAP_000.pdf